CLINICAL TRIAL: NCT07386132
Title: Effect of Position on Ankle Dorsiflexor, Hallux Dorsiflexor and Plantar Flexor Muscle Strength
Brief Title: Effect of Position on Ankle Dorsiflexor, Hallux Dorsiflexor and Plantar Flexor Muscle Strength: Are Ankle Dorsiflexor and Plantar Flexor Muscle Strengths Greater in the Standing Position Compared to the Supine Position?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, deniz erdem yıldız, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-59
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ankle Dorsiflexor, Hallux Dorsiflexor and Plantar Flexor Strength
Keywords: Foot biomechanics, muscle strength, dorsiflexion, plantar flexion, hallux dorsiflexion, positional assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine Position (Experimental): Ankle dorsiflexor , hallux dorsiflexor and plantar flexor muscle strength assessed in the supine position.
  Interventions: Other: Body Position During Muscle Strength Assessment
- Standing Position (Experimental): Ankle dorsiflexor, hallux dorsiflexor and plantar flexor muscle strength assessed in the standing position.
  Interventions: Other: Body Position During Muscle Strength Assessment

INTERVENTIONS:
Other: Body Position During Muscle Strength Assessment — Muscle strength was assessed in both supine and standing positions using standardized isometric testing. The order of testing positions and movement directions was randomized, and no visual feedback of force output was provided to participants.

SUMMARY:
The purpose of this study is to investigate whether there is a difference in ankle dorsiflexor, hallux dorsiflexion and plantar flexor muscle strength measured in the supine position compared with the standing position. Muscle strength assessments are commonly performed in different body positions; however, the effect of weight-bearing and postural demands on ankle muscle strength measurements remains unclear. Understanding the influence of testing position may improve the standardization and clinical interpretation of muscle strength assessments.

DETAILED DESCRIPTION:
Ankle dorsiflexor and plantar flexor muscles play a crucial role in gait, balance, and postural control. Muscle strength measurements of these muscle groups are widely used in both clinical practice and research to evaluate functional capacity and rehabilitation outcomes. Traditionally, strength assessments are performed in non-weight-bearing positions such as supine; however, standing assessments may better reflect functional and postural demands due to the involvement of balance control and weight-bearing.

In this study, ankle dorsiflexor, hallux dorsiflexion and plantar flexor muscle strength will be assessed in both supine and standing positions using standardized measurement procedures. Measurements will be performed under controlled conditions to minimize variability related to posture, stabilization, and examiner influence. The primary objective is to compare muscle strength values obtained in the two positions and to determine whether standing assessments yield significantly different results compared with supine assessments.

The findings of this study are expected to contribute to the optimization of clinical muscle strength evaluation protocols and to provide insight into the role of functional loading and postural control in ankle muscle strength measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 years and older
* No history or clinical diagnosis of lumbar disc herniation
* Ability to stand independently and perform isometric muscle strength testing
* Voluntary participation with written informed consent

Exclusion Criteria:

* History or clinical diagnosis of lumbar disc herniation
* Professional or elite athletes
* History of lower extremity surgery or neurological disease affecting muscle strength
* Acute musculoskeletal injury at the time of assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Isometric Ankle Muscle Strength | Day 1 ( Single assessment session)
  maximum voluntary isometric contraction force of ankle dorsiflexor and plantar flexor muscles measured in supine and standing positions using a custom made force plate

SECONDARY OUTCOMES:
Isometric Hallux Dorsiflexion Strength | Day 1 ( Single assessment session)
  Maximum voluntary isometric contraction force of the hallux dorsiflexor muscles measured in supine and standing positions using a custom made force plate

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine And Rehabilitation Training And Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)